CLINICAL TRIAL: NCT02547428
Title: A Phase 2b, Randomized, Double-Blind, Multicenter, Placebo-Controlled, Crossover, Safety and Efficacy Study of Centanafadine Sustained-Release (CTN SR) in Adults With Attention-Deficit Hyperactivity Disorder (ADHD)
Brief Title: Safety and Efficacy Study of Centanafadine Sustained-Release (CTN SR) in Adults With Attention-Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NVI-EB-1020-202
Record Dates: First submitted 2015-09-08; First posted 2015-09-11 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: centanafadine sustained-release; Attention-Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CTN SR First, Then Placebo (Experimental): Participants received CTN SR tablets starting at a dose of 100 or 200 milligrams (mg) on Day 1. Dose was up titrated up to 800 mg daily dose for up to 3 weeks in Period 1. The dose was decreased based on safety and tolerability based on Investigator's discretion, followed by a washout Period of 1 week followed by matching-placebo for up to 3 weeks in Period 2. The most common total daily dose (TDD) was 400 mg/day.
  Interventions: Drug: CTN SR; Drug: Matching placebo
- Placebo First, Then CTN SR (Experimental): Participants received matching-placebo for up to 3 weeks in Period 1, followed by a washout Period of 1 week, followed by CTN SR tablets starting at a dose of 100 or 200 mg on Day 1. Dose was up titrated up to 800 mg daily dose for up to 3 weeks in Period 2. The dose was decreased based on safety and tolerability based on Investigator's discretion. The most common TDD was 400 mg/day.
  Interventions: Drug: CTN SR; Drug: Matching placebo

INTERVENTIONS:
Drug: CTN SR — CTN SR tablets, daily, Orally.
  Other Names: Centanafadine Sustained-Release
Drug: Matching placebo — Matching-placebo tablets daily, orally.

SUMMARY:
This was a Phase 2b, randomized, double-blind, multicenter, 2-period, 2-treatment, crossover study to evaluate safety and efficacy of CTN SR compared with placebo in adults with ADHD. Efficacy was also evaluated in the subgroup of adults with ADHD treated with a target CTN SR dose of 400 mg/day.

ELIGIBILITY:
Inclusion Criteria:

1. Participant was 18 to 60 years of age, inclusive, at the time of consent.
2. Participant meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD, defined as, established by a comprehensive psychiatric evaluation based on DSM-5 criteria with at least 5 of the 9 subtype criteria met, as determined by the Conners' Adult ADHD Diagnostic Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-4). Note: DSM-5 was used for screening / diagnosis and DSM-4 was used for evaluation throughout the study.
3. Participant had a Baseline score of greater than or equal to 28 using the Attention-Deficit Hyperactivity Disorder Rating Scale IV (ADHD-RS-IV).
4. Participant had a minimum score of 4 on the Clinical Global Impression of Severity at Baseline.
5. Participant was functioning at an age-appropriate level intellectually, as judged by the Investigator.

Exclusion Criteria:

1. Participant had a current comorbid psychiatric disorder that was either controlled with medications prohibited in this study or was uncontrolled and associated with significant symptoms. Exclusionary conditions included any severe comorbid Axis II disorder or severe Axis I disorder (such as post-traumatic stress disorder, psychosis, bipolar illness, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder) or other symptomatic manifestations that, in the opinion of the examining physician, would have contraindicated CTN SR treatment or confound efficacy or safety assessments. Specifically, participants with mild to moderate forms of Axis I disorders (for example, social phobia and dysthymia) may have been included, whereas participants with a lifetime history of psychosis or bipolar disorder were excluded. Comorbid psychiatric diagnosis was established by a Semi-Structured Clinical Interview for DSM-5 Axis I Disorders (the Mini lnternational Neuropsychiatric lnterview, Version 6.0 [M.I.N.I. 6.0]).
2. Participants who were currently considered a suicide risk, any participant who had previously made a suicide attempt, or those who were currently demonstrating active suicidal ideation as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening, or if in the opinion of the investigator the participant was considered a suicide risk. Participants who developed suicidal ideation or behavior during the study as measured by the C-SSRS were discontinued and followed appropriately.
3. The participant had a body mass index of less than 18.5 or greater than or equal to 40 at Baseline.
4. Participant had a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might have confounded the results of safety assessments administered in the study or that might have increased risk to the participant.
5. Participant had a history of seizures (other than infantile febrile seizures), any tic disorder (except transient tic disorder and participant had no episodes greater than or equal to 1 year), or a current diagnosis and/or a known family history of Tourette's Disorder (that is, first degree relatives).
6. Participant had a known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, transient ischemic attack or stroke or other serious cardiac problems that may have placed them at increased vulnerability to potential sympathomimetic effects.
7. Participant had a known family history of sudden cardiac death or ventricular arrhythmia.
8. Participant had a history of significant bleeding or coagulation disorder and/or low platelet levels (less than 130 x 10^9/liter) or increased international normalized ratio (greater than 1.3) at Screening.
9. Participant had a history of cancer (other than noncomplicated basal or squamous cell cancer).
10. Participant had any clinically significant 12-lead electrocardiogram or clinically significant laboratory abnormality at Screening and/or Baseline.
11. Participant had current abnormal thyroid function, as defined as abnormal Screening thyroid stimulating hormone (less than 0.34 or greater than 5.6 micro-International Units/milliliter). Treatment with a stable dose of thyroid medication for at least 3 months was permitted.
12. Participant had a resting sitting systolic blood pressure (SBP) greater than or equal to 140 millimeters of mercury (mm Hg) or diastolic blood pressure (DBP) greater than or equal to 90 mm Hg. No more than 1 repeat measurement was permitted.
13. Participant had a history of hyponatremia.
14. Participant was on an antihypertensive medication of any kind.
15. Participant has a known history of orthostatic hypotension or has an orthostatic blood pressure drop of greater than or equal to 20 mm Hg (based on the drop between sitting and standing [3 minutes] SBP) at Screening or Baseline.
16. Participant had a known history of hypertension.
17. Participant exhibited lifestyle that may have been confounding to safety or efficacy assessments per the judgment of the investigator (for example, exercises, diets or travels extensively).
18. Participant had a known history of glaucoma.
19. Participant had failed to respond to 1 or more adequate courses (for example, adequate dose and duration with poor response as judged by the Investigator) of stimulant therapy.
20. Participant had a recent history (within the past 6 months) of suspected substance abuse or dependence disorder (excluding nicotine) in accordance with DSM-5 criteria.
21. Participant was taking other medications that have central nervous system effects or affected performance, such as sedating antihistamines and decongestant sympathomimetic, or was recently on monoamine oxidase inhibitors (during or within 14 days of investigational product administration). Stable use of bronchodilator inhalers was not exclusionary. This also included use of any psychoactive prescription medication 30 days prior to Screening or psychoactive over-the-counter ) medication or herbal products that required more than a 7-day washout. Participants currently treated with methylphenidate or amphetamine products were permitted and underwent a 7-day washout period. Participants who had taken atomoxetine were required to undergo a 30-day washout.
22. Participant required the frequent or regular use of aspirin, ibuprofen, and naproxen sodium, or is on any anticoagulant, such as warfarin.
23. Participant was taking known potent inhibitors or inducers of common cytochrome P450 enzymes, including herbal products.
24. Participant had a positive urine drug screen (UDS) result at Screening or Baseline. Note: The UDS must be negative at Screening (with the exception of the participant's current ADHD psychostimulant, if applicable) or Baseline, if applicable, for the participant to potentially have been eligible for study participation. The Investigator, in conjunction with the Medical Monitor, evaluated the potential impact of a positive UDS regarding the continued participation of the participant.
25. Participant had taken an investigational product or taken part in a clinical study within 30 days prior to Screening.
26. Investigational site personnel were not permitted to participate in the study.
27. Participant had participated previously in a CTN investigational study.
28. The female participant was pregnant or lactating.
29. Participant had a documented allergy, hypersensitivity, or intolerance to CTN or to any excipients in the reference product.
30. Participant had a history of allergy or hypersensitivity to medications (for example., monoamine reuptake inhibitors or antibiotics).
31. Participant did not agree to or was unable to abstain from consuming alcohol during the study.

    Reproductive Potential Requirements
32. All female participants were required to have a negative serum beta human chorionic gonadotropin pregnancy test at Screening, a negative urine pregnancy test at Baseline, and be either postmenopausal (12 consecutive months of spontaneous amenorrhea and greater than or equal to 51 years of age), surgically sterile and at least 6 weeks post-sterilization or, for females of childbearing potential, had a negative pregnancy test prior to entering the study and agreed to use acceptable methods of contraception.

    Contraceptive Requirements
33. Condoms were to be used with all forms of contraception (that is., double-barrier method). Acceptable contraceptives included the following:

    1. Intrauterine devices
    2. Hormonal contraceptives (oral, depot, patch, injectable, or vaginal ring)
    3. Diaphragms with spermicidal gel or foam
34. Females of childbearing potential were advised to use acceptable contraceptives from the date of informed consent throughout the study period and for the defined follow-up period.
35. If hormonal contraceptives were used, they were to be administered according to the package insert.
36. Females of childbearing potential who were not currently sexually active agreed to use acceptable contraception, as defined above, if they became sexually active during their study participation and for the defined follow-up time period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2016-06-04 (Actual); Study Completion 2016-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Newport Beach, California
  - Bradenton, Florida
  - Maitland, Florida
  - Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 4 sites in United States from 03 Aug 2015 to 4 Jun 2016.
Pre-assignment Details: A total of 85 participants were enrolled in this study. Participants were randomly assigned to 1 of 2 treatment sequences to receive Centanafadine sustained-release (CTN SR) or placebo in sequence 1, followed by washout, followed by crossover treatment with placebo or CTN SR in sequence 2, with each treatment sequence lasting 3 weeks.
Period: Period 1- Treatment Sequence 1 (3 Weeks)
Arm/Group | CTN SR First, Then Placebo | Placebo First, Then CTN SR
Started | 42 | 43
Received at Least 1 Dose of Study Drug | 42 | 43
Completed | 31 | 37
Not Completed | 11 | 6
Not completed — Adverse Event | 8 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Dosing Suspension | 1 | 3
Period: Period 2- Treatment Sequence 2 (3 Weeks)
Arm/Group | CTN SR First, Then Placebo | Placebo First, Then CTN SR
Started | 31 | 37
Completed | 30 | 30
Not Completed | 1 | 7
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Investigator Discretion | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized and had at least one post-dose efficacy assessment.
Groups:
- CTN SR First, Then Placebo: Participants received CTN SR tablets starting at a dose of 100 or 200 mg on Day 1. Dose was up titrated up to 800 mg daily dose for up to 3 weeks in Period 1. The dose was decreased based on safety and tolerability based on Investigator's discretion, followed by a washout Period of 1 week followed by matching-placebo for up to 3 weeks in Period 2. The most common TDD was 400 mg/day.
- Total: Total of all reporting groups
Arm/Group | CTN SR First, Then Placebo | Placebo First, Then CTN SR | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (11.7) | 36.5 (11.9) | 35.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 24 | 24 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 11 | 26
  Not Hispanic or Latino | 27 | 32 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Black or African American | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 28 | 31 | 59
  Multiple | 3 | 1 | 4
  Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Attention-Deficit Hyperactivity Disorder Rating Scale IV (ADHD-RS-IV) Score
Description: The ADHD-RS-IV consists of 18 items and is designed to reflect the participant's current ADHD symptomatology; the severity, frequency, and impairment are measured for each of the items. The 18 items are grouped into 2 subscales of 9 symptoms each: Hyperactivity/Impulsivity (even numbered items 2-18) and Inattentiveness (odd numbered items 1-17). Each item is scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms), with the total score for the rating scale ranging from 0 to 54. Higher scores indicate more severe disease. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 3
Population: FAS Full Analysis Set (FAS) included all participants who were randomized and had at least one post-dose efficacy assessment. Number analyzed is the number of participants with data available for analyses at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CTN SR: Participants received CTN SR tablets starting at a dose of 100 or 200 mg on Day 1. Dose was up titrated up to 800 mg daily dose for up to 3 weeks. The dose was decreased based on safety and tolerability based on Investigator's discretion. The most common total daily dose TDD was 400 mg/day.
- Placebo: Participants received matching-placebo for up to 3 weeks. Placebo was titrated in the same manner to protect the blind. The most common TDD was 400 mg/day.
Arm/Group | CTN SR | Placebo
Number analyzed (Participants) | 85 | 85
score on a scale | -16.2 (11.1) | -7.9 (7.9)
Statistical Analysis 1: Comparison: CTN SR vs Placebo; Null hypothesis was that there was no difference in ADHD-RS-IV total score change from Baseline between CTN SR and placebo. The analysis of covariance (ANCOVA) model included terms for period, sequence, and treatment as fixed effects, and Baseline score as a covariate, and a participate-within-sequence term as a random effect; Test type: Superiority; p < 0.001, ANCOVA; Treatment difference = -8.1, 95% CI 2-sided [-11.0 to -5.1], Standard Error of Mean 1.48 — Sample size of 60 participants (30 per treatment sequence) was needed to provide minimum 85% power to detect 5 point difference between treatments at a 2-sided significance level of 5% using a paired t-test

2. Primary Outcome: Change From Baseline in ADHD-RS-IV Score for Subgroup of Participants With Target CTN SR Dose of 400 mg/Day
Description: as for outcome 1
Time Frame: Baseline and Week 3
Population: FAS included all participants who were randomized and had at least one post-dose efficacy assessment. Overall number analyzed is the number of participants available for analyses. Number analyzed is the number of participants with data available for analyses at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CTN SR 400 mg: Participants received CTN SR 400 mg tablets daily for 3 weeks in treatment Periods 1 and 2.
- Placebo: Participants received matching-placebo daily for 3 weeks in treatment Periods 1 and 2.
Arm/Group | CTN SR 400 mg | Placebo
Number analyzed (Participants) | 47 | 47
score on a scale | -16.3 (11.1) | -8.4 (8.1)
Statistical Analysis 1: Comparison: CTN SR 400 mg vs Placebo; Null hypothesis was that there was no difference in ADHD-RS-IV total score change from Baseline between CTN SR 400 mg/day and placebo; Test type: Superiority; p < 0.001, ANCOVA; Treatment difference = -7.1, 95% CI 2-sided [-10.7 to -3.6], Standard Error of Mean 1.74

3. Secondary Outcome: Change From Baseline in ADHD-RS-IV Score Total Score After 1 and 2 Weeks of Double-blind Treatment
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, and 2
Population: FAS included all participants who were randomized and had at least one post-dose efficacy assessment. Number analyzed is the number of participants with data available for analyses at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CTN SR | Placebo
Number analyzed (Participants) | 85 | 85
score on a scale
  Change from Baseline at Week 1: number analyzed (Participants) | 79 | 74
  Change from Baseline at Week 1 | -12.0 (10.3) | -6.6 (7.7)
  Change from Baseline at Week 2: number analyzed (Participants) | 79 | 74
  Change from Baseline at Week 2 | -15.4 (10.6) | -7.6 (7.9)

4. Secondary Outcome: Change From Baseline in ADHD-RS-IV Score Total Score After 1 and 2 Weeks of Double-blind Treatment for Subgroup of Participants With Target CTN SR Dose of 400 mg/Day
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, and 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CTN SR 400 mg | Placebo
Number analyzed (Participants) | 47 | 47
score on a scale
  Change from Baseline at Week 1: number analyzed (Participants) | 45 | 46
  Change from Baseline at Week 1 | -12.0 (10.1) | -7.7 (8.5)
  Change from Baseline at Week 2: number analyzed (Participants) | 45 | 46
  Change from Baseline at Week 2 | -15.0 (10.4) | -8.3 (8.2)

5. Secondary Outcome: Change From Baseline in ADHD-RS-IV Inattention Subscale Score of Double-blind Treatment
Description: The ADHD-RS-IV consists of 18 items and is designed to reflect the participant's current ADHD symptomatology; the severity, frequency, and impairment are measured for each of the items. The 18 items are grouped into 2 subscales of 9 symptoms each: Hyperactivity/Impulsivity (even numbered items 2-18) and Inattentiveness (odd numbered items 1-17). Each item is scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms), with the total score for the rating scale ranging from 0 to 54. The possible sub-scale score range is from 0 to 27. Higher scores indicate more severe disease. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 1, 2 and 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CTN SR | Placebo
Number analyzed (Participants) | 85 | 85
score on a scale
  Change from Baseline at Week 1: number analyzed (Participants) | 79 | 74
  Change from Baseline at Week 1 | -7.0 (6.2) | -3.6 (4.6)
  Change from Baseline at Week 2: number analyzed (Participants) | 79 | 74
  Change from Baseline at Week 2 | -9.2 (6.7) | -4.2 (5.0)
  Change from Baseline at Week 3: number analyzed (Participants) | 79 | 74
  Change from Baseline at Week 3 | -9.3 (6.8) | -4.3 (5.2)

6. Secondary Outcome: Change From Baseline in ADHD-RS-IV Inattention Subscale Score of Double-blind Treatment for Subgroup of Participants With Target CTN SR Dose of 400 mg/Day
Description: as for outcome 5
Time Frame: Baseline, Weeks 1, 2 and 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CTN SR 400 mg | Placebo
Number analyzed (Participants) | 47 | 47
score on a scale
  Change from Baseline at Week 1: number analyzed (Participants) | 45 | 46
  Change from Baseline at Week 1 | -6.6 (6.2) | -4.5 (5.1)
  Change from Baseline at Week 2: number analyzed (Participants) | 45 | 46
  Change from Baseline at Week 2 | -9.4 (6.7) | -4.8 (5.0)
  Change from Baseline at Week 3: number analyzed (Participants) | 45 | 46
  Change from Baseline at Week 3 | -9.7 (6.7) | -4.8 (5.2)

7. Secondary Outcome: Change From Baseline in ADHD-RS-IV Hyperactivity/Impulsivity Subscale Score of Double-blind Treatment
Description: as for outcome 5
Time Frame: Baseline, Weeks 1, 2 and 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CTN SR | Placebo
Number analyzed (Participants) | 85 | 85
score on a scale
  Change from Baseline at Week 1: number analyzed (Participants) | 79 | 74
  Change from Baseline at Week 1 | -5.0 (5.8) | -2.9 (4.5)
  Change from Baseline at Week 2: number analyzed (Participants) | 79 | 74
  Change from Baseline at Week 2 | -6.2 (5.7) | -3.4 (4.6)
  Change from Baseline at Week 3: number analyzed (Participants) | 79 | 74
  Change from Baseline at Week 3 | -6.9 (6.0) | -3.6 (4.7)

8. Secondary Outcome: Change From Baseline in ADHD-RS-IV Hyperactivity/Impulsivity Subscale Score of Double-blind Treatment for Subgroup of Participants With Target CTN SR Dose of 400 mg/Day
Description: as for outcome 5
Time Frame: Baseline, Weeks 1, 2 and 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CTN SR 400 mg | Placebo
Number analyzed (Participants) | 47 | 47
score on a scale
  Change from Baseline at Week 1: number analyzed (Participants) | 45 | 46
  Change from Baseline at Week 1 | -5.3 (6.1) | -3.2 (5.0)
  Change from Baseline at Week 2: number analyzed (Participants) | 45 | 46
  Change from Baseline at Week 2 | -5.6 (5.5) | -3.5 (5.0)
  Change from Baseline at Week 3: number analyzed (Participants) | 45 | 46
  Change from Baseline at Week 3 | -6.6 (6.1) | -3.6 (5.2)

9. Secondary Outcome: Permanent Product Measure of Performance (PERMP) Score
Description: The Permanent Product Measure of Performance (PERMP) is a skill-adjusted math test consisting of 400 problems. The PERMP total score is the sum of the number of math problems attempted plus the number of math problems answered correctly in a 10-minute session. The score range of number of math problems attempted and number of math problems answered correctly is 0-400 and the total score range from 0-800. The higher scores indicate better performance. Higher scores mean higher performance and less severe ADHD symptoms.
Time Frame: Predose -0.5 hour and post-dose 1, 3, 5, 7, 9, 11 and 13 hours at Weeks 4 and 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CTN SR | Placebo
Number analyzed (Participants) | 58 | 58
score on a scale
  Total Score- 0.5 Hour Before Dosing | 226.7 (87.1) | 232.7 (90.9)
  Total Score- 1 Hour After Dosing | 238.7 (90.4) | 246.2 (94.4)
  Total Score- 3 Hour After Dosing: number analyzed (Participants) | 57 | 58
  Total Score- 3 Hour After Dosing | 246.2 (96.3) | 242.6 (94.4)
  Total Score- 5 Hour After Dosing: number analyzed (Participants) | 57 | 58
  Total Score- 5 Hour After Dosing | 244.5 (92.2) | 246.0 (95.3)
  Total Score- 7 Hour After Dosing: number analyzed (Participants) | 57 | 58
  Total Score- 7 Hour After Dosing | 244.6 (95.3) | 245.8 (100.1)
  Total Score- 9 Hour After Dosing: number analyzed (Participants) | 57 | 57
  Total Score- 9 Hour After Dosing | 246.6 (91.1) | 245.4 (99.5)
  Total Score- 11 Hour After Dosing: number analyzed (Participants) | 58 | 57
  Total Score- 11 Hour After Dosing | 250.9 (91.5) | 244.9 (104.5)
  Total Score- 13 Hour After Dosing: number analyzed (Participants) | 58 | 57
  Total Score- 13 Hour After Dosing | 250.7 (93.5) | 244.0 (101.4)
  Number of Math Problems Attempted- 0.5 Hour Before Dosing | 115.3 (43.5) | 119.0 (45.6)
  Number of Math Problems Attempted- 1 Hour After Dosing | 121.3 (45.3) | 126.1 (47.6)
  Number of Math Problems Attempted- 3 Hour After Dosing: number analyzed (Participants) | 57 | 58
  Number of Math Problems Attempted- 3 Hour After Dosing | 124.9 (48.3) | 123.8 (47.8)
  Number of Math Problems Attempted- 5 Hour After Dosing: number analyzed (Participants) | 57 | 58
  Number of Math Problems Attempted- 5 Hour After Dosing | 124.2 (46.4) | 125.7 (47.9)
  Number of Math Problems Attempted- 7 Hour After Dosing: number analyzed (Participants) | 57 | 58
  Number of Math Problems Attempted- 7 Hour After Dosing | 124.2 (47.9) | 125.4 (50.4)
  Number of Math Problems Attempted- 9 Hour After Dosing: number analyzed (Participants) | 57 | 57
  Number of Math Problems Attempted- 9 Hour After Dosing | 125.0 (45.6) | 125.2 (50.1)
  Number of Math Problems Attempted- 11 Hour After Dosing: number analyzed (Participants) | 58 | 57
  Number of Math Problems Attempted- 11 Hour After Dosing | 127.2 (45.7) | 124.2 (52.5)
  Number of Math Problems Attempted- 13 Hour After Dosing: number analyzed (Participants) | 58 | 57
  Number of Math Problems Attempted- 13 Hour After Dosing | 127.1 (46.8) | 124.0 (51.0)
  Number of Math Problems Answered Correctly- 0.5 Hour Before Dosing | 111.4 (43.7) | 113.7 (45.8)
  Number of Math Problems Answered Correctly- 1 Hour After Dosing | 117.3 (45.2) | 120.1 (47.5)
  Number of Math Problems Answered Correctly- 3 Hour After Dosing: number analyzed (Participants) | 57 | 58
  Number of Math Problems Answered Correctly- 3 Hour After Dosing | 121.3 (48.1) | 118.8 (47.2)
  Number of Math Problems Answered Correctly- 5 Hour After Dosing: number analyzed (Participants) | 57 | 58
  Number of Math Problems Answered Correctly- 5 Hour After Dosing | 120.3 (45.9) | 120.3 (48.0)
  Number of Math Problems Answered Correctly- 7 Hour After Dosing: number analyzed (Participants) | 57 | 58
  Number of Math Problems Answered Correctly- 7 Hour After Dosing | 120.4 (47.5) | 120.4 (50.2)
  Number of Math Problems Answered Correctly- 9 Hour After Dosing: number analyzed (Participants) | 57 | 57
  Number of Math Problems Answered Correctly- 9 Hour After Dosing | 121.6 (45.6) | 120.2 (49.9)
  Number of Math Problems Answered Correctly- 11 Hour After Dosing: number analyzed (Participants) | 58 | 57
  Number of Math Problems Answered Correctly- 11 Hour After Dosing | 123.7 (45.8) | 120.6 (52.1)
  Number of Math Problems Answered Correctly- 13 Hour After Dosing: number analyzed (Participants) | 58 | 57
  Number of Math Problems Answered Correctly- 13 Hour After Dosing | 123.6 (46.8) | 120.0 (50.5)

10. Secondary Outcome: PERMP Score for Subgroup of Participants With Target CTN SR Dose of 400 mg/Day
Description: The PERMP is a skill-adjusted math test consisting of 400 problems. The PERMP total score is the sum of the number of math problems attempted plus the number of math problems answered correctly in a 10-minute session. The score range of number of math problems attempted and number of math problems answered correctly is 0-400 and the total score range from 0-800. The higher scores indicate better performance. Higher scores mean higher performance and less severe ADHD symptoms.
Time Frame: Predose -0.5 hour and post-dose 1, 3, 5, 7, 9, 11 and 13 hours at Weeks 4 and 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CTN SR 400 mg | Placebo
Number analyzed (Participants) | 47 | 47
score on a scale
  Total Score- 0.5 Hour Before Dosing: number analyzed (Participants) | 42 | 41
  Total Score- 0.5 Hour Before Dosing | 226.8 (81.4) | 229.1 (88.4)
  Total Score- 1 Hour After Dosing: number analyzed (Participants) | 42 | 41
  Total Score- 1 Hour After Dosing | 241.5 (82.1) | 242.6 (89.1)
  Total Score- 3 Hour After Dosing: number analyzed (Participants) | 41 | 41
  Total Score- 3 Hour After Dosing | 249.8 (90.0) | 240.4 (94.4)
  Total Score- 5 Hour After Dosing: number analyzed (Participants) | 41 | 41
  Total Score- 5 Hour After Dosing | 248.8 (88.0) | 241.0 (95.3)
  Total Score- 7 Hour After Dosing: number analyzed (Participants) | 41 | 41
  Total Score- 7 Hour After Dosing | 249.7 (96.2) | 245.6 (96.6)
  Total Score- 9 Hour After Dosing: number analyzed (Participants) | 41 | 40
  Total Score- 9 Hour After Dosing | 249.5 (88.7) | 246.2 (98.9)
  Total Score- 11 Hour After Dosing: number analyzed (Participants) | 42 | 40
  Total Score- 11 Hour After Dosing | 253.5 (91.8) | 246.1 (102.4)
  Total Score- 13 Hour After Dosing: number analyzed (Participants) | 42 | 40
  Total Score- 13 Hour After Dosing | 257.5 (96.9) | 248.6 (96.5)
  Number of Math Problems Attempted- 0.5 Hour Before Dosing: number analyzed (Participants) | 42 | 41
  Number of Math Problems Attempted- 0.5 Hour Before Dosing | 115.4 (40.6) | 116.6 (44.2)
  Number of Math Problems Attempted- 1 Hour After Dosing: number analyzed (Participants) | 42 | 41
  Number of Math Problems Attempted- 1 Hour After Dosing | 122.9 (40.9) | 123.4 (44.8)
  Number of Math Problems Attempted- 3 Hour After Dosing: number analyzed (Participants) | 41 | 41
  Number of Math Problems Attempted- 3 Hour After Dosing | 127.0 (45.0) | 122.2 (47.8)
  Number of Math Problems Attempted- 5 Hour After Dosing: number analyzed (Participants) | 41 | 41
  Number of Math Problems Attempted- 5 Hour After Dosing | 126.4 (44.2) | 122.5 (47.6)
  Number of Math Problems Attempted- 7 Hour After Dosing: number analyzed (Participants) | 41 | 41
  Number of Math Problems Attempted- 7 Hour After Dosing | 126.9 (48.2) | 124.6 (48.5)
  Number of Math Problems Attempted- 9 Hour After Dosing: number analyzed (Participants) | 41 | 40
  Number of Math Problems Attempted- 9 Hour After Dosing | 126.6 (44.3) | 125.0 (49.4)
  Number of Math Problems Attempted- 11 Hour After Dosing: number analyzed (Participants) | 42 | 40
  Number of Math Problems Attempted- 11 Hour After Dosing | 128.6 (45.8) | 124.6 (51.2)
  Number of Math Problems Attempted- 13 Hour After Dosing: number analyzed (Participants) | 42 | 40
  Number of Math Problems Attempted- 13 Hour After Dosing | 130.4 (48.5) | 126.1 (48.4)
  Number of Math Problems Answered Correctly- 0.5 Hour Before Dosing: number analyzed (Participants) | 42 | 41
  Number of Math Problems Answered Correctly- 0.5 Hour Before Dosing | 111.4 (41.0) | 112.6 (44.3)
  Number of Math Problems Answered Correctly- 1 Hour After Dosing: number analyzed (Participants) | 42 | 41
  Number of Math Problems Answered Correctly- 1 Hour After Dosing | 118.6 (41.3) | 119.2 (44.4)
  Number of Math Problems Answered Correctly- 3 Hour After Dosing: number analyzed (Participants) | 41 | 41
  Number of Math Problems Answered Correctly- 3 Hour After Dosing | 122.9 (45.1) | 118.3 (46.7)
  Number of Math Problems Answered Correctly- 5 Hour After Dosing: number analyzed (Participants) | 41 | 41
  Number of Math Problems Answered Correctly- 5 Hour After Dosing | 122.4 (43.9) | 118.6 (47.8)
  Number of Math Problems Answered Correctly- 7 Hour After Dosing: number analyzed (Participants) | 41 | 41
  Number of Math Problems Answered Correctly- 7 Hour After Dosing | 122.9 (48.0) | 121.0 (48.2)
  Number of Math Problems Answered Correctly- 9 Hour After Dosing: number analyzed (Participants) | 41 | 40
  Number of Math Problems Answered Correctly- 9 Hour After Dosing | 122.9 (44.5) | 121.2 (49.6)
  Number of Math Problems Answered Correctly- 11 Hour After Dosing: number analyzed (Participants) | 42 | 40
  Number of Math Problems Answered Correctly- 11 Hour After Dosing | 124.9 (46.1) | 121.5 (51.3)
  Number of Math Problems Answered Correctly- 13 Hour After Dosing: number analyzed (Participants) | 42 | 40
  Number of Math Problems Answered Correctly- 13 Hour After Dosing | 127.1 (48.5) | 122.5 (48.1)

11. Secondary Outcome: Number of Participants With Clinical Global Impressions of Severity (CGI-S) Score
Description: The CGI-S is performed to rate the severity of a participant's condition on a 8- point scale ranging from 0 to 7 where 0=not assessed, 1=normal, not at all ill, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7 = among the most extremely ill participants.
Time Frame: Baseline
Population: FAS included all participants who were randomized and had at least one post-dose efficacy assessment. The data is reported as per the crossover dose received.
Measure: Count of Participants; unit: Participants
Arm/Group | CTN SR First, Then Placebo | Placebo First, Then CTN SR
Number analyzed (Participants) | 42 | 43
Participants
  Moderately ill | 22 | 18
  Markedly ill | 15 | 22
  Severely ill | 5 | 3

12. Secondary Outcome: Number of Participants With Clinical Global Impressions of Improvement (CGI-I) Score
Description: The CGI-I permits a global evaluation of the participant's improvement over time. The CGI-I is a 8-point scale ranging from 0 to 7 where 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse and 7=very much worse. The CGI-I is completed by the clinician and assesses the participant's improvement relative to the symptoms at Baseline.
Time Frame: Weeks 1, 2, and 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CTN SR | Placebo
Number analyzed (Participants) | 85 | 85
Participants
  Week 1: number analyzed (Participants) | 68 | 68
  Week 1: Score 1 | 4 | 0
  Week 1: Score 2 | 19 | 8
  Week 1: Score 3 | 22 | 19
  Week 1: Score 4 | 22 | 41
  Week 1: Score 5 | 1 | 0
  Week 1: Score 6 | 0 | 0
  Week 1: Score 7 | 0 | 0
  Week 2: number analyzed (Participants) | 68 | 68
  Week 2: Score 1 | 16 | 2
  Week 2: Score 2 | 17 | 9
  Week 2: Score 3 | 19 | 17
  Week 2: Score 4 | 16 | 39
  Week 2: Score 5 | 0 | 1
  Week 2: Score 6 | 0 | 0
  Week 2: Score 7 | 0 | 0
  Week 3: number analyzed (Participants) | 68 | 68
  Week 3: Score 1 | 16 | 2
  Week 3: Score 2 | 18 | 8
  Week 3: Score 3 | 19 | 21
  Week 3: Score 4 | 15 | 37
  Week 3: Score 5 | 0 | 0
  Week 3: Score 6 | 0 | 0
  Week 3: Score 7 | 0 | 0

13. Secondary Outcome: Number of Participants With CGI-I Score for Subgroup of Participants With Target CTN SR Dose of 400 mg/Day
Description: as for outcome 12
Time Frame: Weeks 1, 2, and 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | CTN SR 400 mg | Placebo
Number analyzed (Participants) | 47 | 47
Participants
  Week 1: number analyzed (Participants) | 44 | 44
  Week 1: Score 1 | 2 | 0
  Week 1: Score 2 | 11 | 6
  Week 1: Score 3 | 16 | 15
  Week 1: Score 4 | 14 | 23
  Week 1: Score 5 | 1 | 0
  Week 1: Score 6 | 0 | 0
  Week 1: Score 7 | 0 | 0
  Week 2: number analyzed (Participants) | 44 | 44
  Week 2: Score 1 | 8 | 1
  Week 2: Score 2 | 13 | 6
  Week 2: Score 3 | 11 | 11
  Week 2: Score 4 | 12 | 26
  Week 2: Score 5 | 0 | 0
  Week 2: Score 6 | 0 | 0
  Week 2: Score 7 | 0 | 0
  Week 3: number analyzed (Participants) | 44 | 44
  Week 3: Score 1 | 8 | 0
  Week 3: Score 2 | 14 | 6
  Week 3: Score 3 | 14 | 17
  Week 3: Score 4 | 8 | 21
  Week 3: Score 5 | 0 | 0
  Week 3: Score 6 | 0 | 0
  Week 3: Score 7 | 0 | 0

14. Secondary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A TEAE was defined as any AE with onset post study drug treatment in the two crossover treatment periods. As prespecified in the protocol, data for safety is reported by the treatment group (CTN SR and placebo).
Time Frame: From signing of informed consent up to approximately Week 9
Population: Safety population included all participants who were randomized and had taken any dose of investigational product (including placebo) in the Double-blind Crossover Phase.
Measure: Count of Participants; unit: Participants
Arm/Group | CTN SR | Placebo
Number analyzed (Participants) | 79 | 74
Participants | 63 | 50

15. Secondary Outcome: Number of Participants With at Least One TEAEs for Subgroup of Participants With Target CTN SR Dose of 400 mg/Day
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A TEAE was defined as any AE with onset post study drug treatment in the two crossover treatment periods. As prespecified in the protocol, data for safety is reported by the treatment group (CTN SR and placebo).
Time Frame: From signing of informed consent up to approximately Week 9
Population: Safety population included all participants who were randomized and had taken any dose of investigational product (including placebo) in the Double-blind Crossover Phase. Overall number analyzed is the number of participants available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | CTN SR 400 mg | Placebo
Number analyzed (Participants) | 45 | 46
Participants | 32 | 30

16. Secondary Outcome: Cmax: Maximum Concentration
Time Frame: Predose 90 minutes and 2, 4, 6, 8,10, 11 to 12 and 24 hours post-dose at Weeks 4 and 8
Population: The Pharmacokinetic Analysis Set included all participants in the Safety Population who have post-dose drug concentration data available for analysis. Overall number analyzed is the number of participants available for analyses.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Groups:
- CTN SR 300 mg: Participants received CTN SR 300 mg tablet for up to 3 weeks in treatment Periods 1 and 2.
- CTN SR 400 mg: Participants received CTN SR 400 mg tablet for up to 3 weeks in treatment Periods 1 and 2.
- CTN SR 600 mg: Participants received CTN SR 600 mg tablet for up to 3 weeks in treatment Periods 1 and 2.
Arm/Group | CTN SR 300 mg | CTN SR 400 mg | CTN SR 600 mg
Number analyzed (Participants) | 4 | 33 | 6
nanograms per milliliter (ng/ml) | 1450 (461) | 1460 (570) | 3080 (2260)

17. Secondary Outcome: Tmax: Time to Maximum Concentration
Time Frame: Predose 90 minutes and 2, 4, 6, 8,10, 11 to 12 and 24 hours post-dose at Weeks 4 and 8
Population: as for outcome 16
Measure: Median (Full Range); unit: hour
Arm/Group | CTN SR 300 mg | CTN SR 400 mg | CTN SR 600 mg
Number analyzed (Participants) | 4 | 33 | 6
hour | 3.36 [2.00 to 6.48] | 8.10 [1.95 to 12.0] | 8.12 [1.72 to 11.5]

18. Secondary Outcome: AUC0-t: Area Under the Concentration-Time Curve During the Steady-State 24-hour Dosing Interval
Time Frame: Predose 90 minutes and 2, 4, 6, 8,10, 11 to 12 and 24 hours post-dose at Weeks 4 and 8
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | CTN SR 300 mg | CTN SR 400 mg | CTN SR 600 mg
Number analyzed (Participants) | 4 | 33 | 6
hours*ng/mL | 14700 (5180) | 16900 (5970) | 34300 (23600)

19. Secondary Outcome: t½: Elimination Phase Half-Life
Time Frame: Predose 90 minutes and 2, 4, 6, 8,10, 11 to 12 and 24 hours post-dose at Weeks 4 and 8
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | CTN SR 300 mg | CTN SR 400 mg | CTN SR 600 mg
Number analyzed (Participants) | 4 | 15 | 5
hour | 5.53 (3.30) | 5.08 (2.88) | 4.06 (1.89)

20. Secondary Outcome: Clast: Last Measurable Concentration
Time Frame: Predose 90 minutes and 2, 4, 6, 8,10, 11 to 12 and 24 hours post-dose at Weeks 4 and 8
Population: All efforts have been exhausted to locate this data and it has since been destroyed, therefore no data is available to report for this outcome measure.
Arm/Group | CTN SR 300 mg | CTN SR 400 mg | CTN SR 600 mg
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Tlast: Time Point of the Last Measurable Concentration
Time Frame: Predose 90 minutes and 2, 4, 6, 8,10, 11 to 12 and 24 hours post-dose at Weeks 4 and 8
Population: as for outcome 20
Arm/Group | CTN SR 300 mg | CTN SR 400 mg | CTN SR 600 mg
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: ke: Elimination Phase Rate Constant
Time Frame: Predose 90 minutes and 2, 4, 6, 8,10, 11 to 12 and 24 hours post-dose at Weeks 4 and 8
Population: as for outcome 20
Arm/Group | CTN SR 300 mg | CTN SR 400 mg | CTN SR 600 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to approximately Week 9
Description: Safety Population consisted of all participants who were randomized and had taken any dose of investigational product in the Double-blind Crossover Phase. As prespecified in the protocol, data for safety is reported by the treatment group (CTN SR and placebo).
Groups:
- CTN SR: Participants received CTN SR tablets at a starting dose of 100 or 200 mg on Day 1. Dose was up titrated up to 800 mg daily dose for up to 3 weeks. The dose was decreased based on safety and tolerability based on Investigator's discretion. The most common TDD was 400 mg/day.
Arm/Group | CTN SR | Placebo
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/74
Other Adverse Events (participants affected / at risk) | 63/79 | 50/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CTN SR (N=79) | Placebo (N=74)
Tachycardia (Cardiac disorders) | 9 | 7
Palpitations (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vision Blurred (Eye disorders) | 3 | 0
Dry Eye (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 16 | 0
Diarrohea (Gastrointestinal disorders) | 14 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Toothache (Gastrointestinal disorders) | 2 | 3
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Discomfort (General disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 1
Food Poisoning (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 11 | 0
Chest Discomfort (General disorders) | 2 | 1
Energy Increased (General disorders) | 1 | 0
Feeling Abnormal (General disorders) | 1 | 0
Sluggishness (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Infusion Site Bruising (General disorders) | 0 | 1
Vessel Puncture Site Haemorrhage (General disorders) | 0 | 1
Vessel Puncture Site Pain (General disorders) | 0 | 1
Choleithiasis (Hepatobiliary disorders) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 7
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1
Tooth Abscess (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 2 | 0
Orthostatic Heart Rate Response Increased (Investigations) | 6 | 0
Blood Pressure Increased (Investigations) | 2 | 1
Hepatic Enzyme Increased (Investigations) | 2 | 0
Weight Decreased (Investigations) | 2 | 0
Blood Pressure Diastolic Increased (Investigations) | 1 | 3
Blood Pressure Orthostatic Decreased (Investigations) | 1 | 0
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1 | 1
Heart Rate Increased (Investigations) | 1 | 0
Liver Function Test Abnormal (Investigations) | 1 | 0
Lymph Node Palpable (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1
Blood Pressure Systolic Increased (Investigations) | 0 | 1
Weight Increased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 19 | 0
Increased Appetite (Metabolism and nutrition disorders) | 2 | 0
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 18 | 6
Dizziness (Nervous system disorders) | 6 | 1
Dysgeusia (Nervous system disorders) | 4 | 0
Poor Quality Sleep (Nervous system disorders) | 2 | 0
Mental Impairment (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 1
Tension Headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 1
Sinus Headache (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 9 | 2
Irritability (Psychiatric disorders) | 4 | 3
Agitation (Psychiatric disorders) | 3 | 0
Affect Lability (Psychiatric disorders) | 2 | 0
Bruxism (Psychiatric disorders) | 2 | 0
Derealisation (Psychiatric disorders) | 2 | 0
Dysphoria (Psychiatric disorders) | 2 | 0
Restlessness (Psychiatric disorders) | 2 | 0
Suicidal Ideation (Psychiatric disorders) | 2 | 0
Abnormal Dreams (Psychiatric disorders) | 1 | 3
Apathy (Psychiatric disorders) | 1 | 0
Emotional Disorder (Psychiatric disorders) | 1 | 0
Jealous Delusion (Psychiatric disorders) | 1 | 0
Libido Decreased (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Pressure Of Speech (Psychiatric disorders) | 1 | 0
Initial Insomnia (Psychiatric disorders) | 0 | 5
Middle Insomnia (Psychiatric disorders) | 0 | 4
Terminal Insomnia (Psychiatric disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 8 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2
Sinus Operation (Surgical and medical procedures) | 0 | 1
Flushing (Vascular disorders) | 2 | 0
Hot Flush (Vascular disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 11 | 0
Infusion Site Pain (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.